CLINICAL TRIAL: NCT05833048
Title: Rectus Sheath Block in Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ali Nima Shariat, Associate Professor of Anesthesiology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-23-00096
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Disease; Postoperative Pain
Keywords: cardiac surgery; regional anesthesia
MeSH Terms: conditions — Heart Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectus Sheath Block (Experimental)
  Interventions: Procedure: Rectus sheath block
- No block (No Intervention)

INTERVENTIONS:
Procedure: Rectus sheath block — Participants will receive an ultrasound guided rectus sheath block with local anesthetic
  Arms: Rectus Sheath Block

SUMMARY:
This is a prospective, randomized study. The purpose of this study is to evaluate the effect of post-surgical pain control of a type of peripheral nerve block, Rectus Sheath Block.

1. Does the rectus sheath block decrease opioid consumption postoperatively after cardiac surgery?
2. Does the rectus sheath block decrease VAS pain scores postoperatively after cardiac surgery? Study participants will be assigned to receive either rectus sheath block or no block.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  1. Adults 18-85 years old
  2. Scheduled to undergo cardiac procedures involving chest tubes
  3. Male or female

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. ASA class V
  2. Urgent or emergent surgery
  3. Contraindications to administration of local anesthesia (e.g. local anesthetic allergy)
  4. History of substance abuse or chronic opioid use
  5. Patient refusal or inability to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 72 hours postoperatively
  Amount of opioid consumption required postoperatively
VAS pain scores | 72 hours postoperatively
  VAS pain scores (1-10, 1 being no pain and 10 being worst pain) recorded postoperatively

SECONDARY OUTCOMES:
Length of stay in ICU | 72 hours
  Amount of time spent in ICU postoperatively
Length of hospital stay | 72 hours
  Length of time spent in hospital postoperatively
Time to extubation | 72 hours
  Length of time requiring postoperative mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Morningside Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No